CLINICAL TRIAL: NCT00945399
Title: Phase III Protocol Comparing a Microfracture Treatment to a CARTIPATCH® Chondrocyte Graft Treatment in Femoral Condyle Lesions
Brief Title: Comparison of Microfracture Treatment and CARTIPATCH® Chondrocyte Graft Treatment in Femoral Condyle Lesions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Manufacturing stopped
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003481-18
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Knee Chondral; Osteochondral Defect
MeSH Terms: interventions — Arthroplasty, Subchondral

ARMS (2):
- Autologous Chondrocytes Implantation (Experimental)
  Interventions: Procedure: CARTIPATCH® procedure
- Microfracture (Active Comparator)
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: CARTIPATCH® procedure — Cartilage is harvested and treated for chondrocytes isolation and culture. After multiplication, the chondrocytes are transferred into a biomaterial support and surgically implanted.
  Arms: Autologous Chondrocytes Implantation
Procedure: Microfracture — Tiny fractures are created at the cartilage surface to stimulate cartilage growth.
  Arms: Microfracture

SUMMARY:
CARTIPATCH® is an Autologous Chondrocyte Implantation product including functional cells in a matrix, indicated for the treatment of isolated osteocartilaginous lesions. The submitted protocol is a Phase III multicentric, prospective, controlled and randomized clinical trial, sponsored by TBF Génie Tissulaire, France. The main objective of the protocol is to compare the clinical improvement of the IKDC subjective score between the microfracture-treated group and the CARTIPATCH® chondrocyte graft-treated group , 18 months following surgery. Several secondary objectives were determined. The microfracture procedure will be conducted in one operative step, during arthroscopy and CARTIPATCH® procedure will be conducted in two operative steps:

1. Arthroscopy to collect cartilage;
2. Implantation following arthrotomy about 6 weeks following arthroscopy.

Both groups will follow the same rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* isolated femoral osteochondral lesion
* aged 18 to 45
* grade 3 or 4 lesion (ICRS) sized 2,5 to 7,5cm2
* lesion depth under 10mm
* IKDC score below 55
* no prior surgical treatment

Exclusion Criteria:

* pregnancy or breastfeeding
* allergy
* arthrosis
* varus or valgus angle greater than 6°
* kissing lesion
* affection of the patella
* excessive laxity
* meniscal pathology history
* severe chronic disease
* BMI > 30
* HIV, Hepatitis B, C, HTLV, Syphilis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation scoring system: IKDC | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gent University Hospital, Dept of Orthopaedic Surgery, Ghent, Belgium